CLINICAL TRIAL: NCT01717677
Title: Preference Based Randomized Trial for Evaluation of Four Treatment Modalities in Prostate Cancer With Low or "Early Intermediate" Risk
Brief Title: Evaluation of Four Treatment Modalities in Prostate Cancer With Low or "Early Intermediate" Risk
Acronym: PREFERE
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Insufficient Recruitment
Sponsor: Association of Urologic Oncology (AUO) (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AP 65/11; DRKS00004405 (Registry Identifier: Freiburger Register)
Record Dates: First submitted 2012-10-26; First posted 2012-10-30 (Estimated); Last update posted 2021-02-10 (Actual); Status verified 2021-02

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Watchful Waiting

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- radical prostatectomy (Experimental): Procedure/Surgery: radical prostatectomy
  Interventions: Procedure: radical prostatectomy
- percutaneous radiation therapy (Experimental): Radiation: percutaneous radiation therapy
  Interventions: Radiation: percutaneous radiation therapy
- permanent seed implantation (Experimental): Radiation: permanent seed implantation
  Interventions: Radiation: permanent seed implantation
- Active Surveillance (Experimental): Procedure/Surgery: Active Surveillance
  Interventions: Procedure: Active Surveillance

INTERVENTIONS:
Procedure: radical prostatectomy
  Arms: radical prostatectomy
Radiation: percutaneous radiation therapy
  Arms: percutaneous radiation therapy
Radiation: permanent seed implantation
  Arms: permanent seed implantation
Procedure: Active Surveillance
  Arms: Active Surveillance

SUMMARY:
4arms preference based Study to compare four therapy options in prostate cancer with low or early intermediate risk

DETAILED DESCRIPTION:
The study will compare four possible therapy options for treatment of newly diagnosed prostate cancer with low or "early intermediate" risk according to the patients preferences.

The Following hypotheses will be tested:

* Radiation is not relevantly worse compared to prostatectomy with regard to time to prostate cancer-related deaths
* Permanent seed implantation therapy not inferior to prostatectomy with regard to time to prostate cancer-related deaths.
* Active Surveillance does not lead to a significant decrease of time to prostate cancer-related deaths compared to prostatectomy.

That for patients with newly diagnosed prostate cancer will be randomized into one of the four treatment arms. Randomization may be limited to at least two of the four treatment arms if a patient refuses one or two of the four treatment arms according to his own preference.

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed, biopsy proven adenocarcinoma of the prostate (ultrasound guided biopsy by standardized protocol)
* Men aged 18-75 years
* Recruitment within 3 months after histological confirmation
* Localized prostata cancer <= cT2a, NX or N0 M0
* PSA <= 10 ng / ml
* Gleason score <= 7a (3 +4)
* ECOG performance status 0 or 1
* <= 30% positive biopsy cores with largest contiguous tumor length <= 5 mm
* IPSS score < 18
* Urine flow (Qmax):> 15 ml / s

Exclusion Criteria:

* Unifocal Gleason 6 cancer <1mm
* History of treatment for BPH e.g. TURP, HIFU or cryotherapy
* History of radiation therapy to the pelvis
* Life expectancy <10 years
* ASA >= 4
* Post-void residual urine > 50 ml
* Prostate volume on transrectal ultrasound > 60 cm3
* large median prostate lobe visualized on transrectal ultrasound
* chronic intestinal inflammatory disease covering the rectum
* Other active malignancy within the past 5 years (except for superficial basal cell carcinoma or non muscle infiltrating bladder carcinoma)
* contraindications for prostatectomy, radiation therapy or Active Surveillance
* Patients refusing written informed consent

Ages: 18 Years to 75 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 457 (Actual)
Dates: Start 2012-10; Primary Completion 2018-01-31 (Actual); Study Completion 2018-04-30 (Actual)

PRIMARY OUTCOMES:
Prostate cancer-specific survival | minimal observation time of 13 years for last study patient

SECONDARY OUTCOMES:
- Overall survival | minimal observation time of 13 years for last study patient
- Time to onset of hormone therapy | 17 years
- Occurrence of the first progression on hormone therapy | 17 years
- Quality of life on EORTC-QLQ-C30 with additional modul PCA (EORTCQLQ- PR25) as well as HADS-D at baseline | before and 3 Mon. after therapy as well as after 1, 2, 3, 5, 7, 10 and 13 years
- Complications / Safety | median 15 years

CONTACTS AND LOCATIONS:
Overall Officials: Michael Stöckle, Prof. Dr., Principal Investigator — Klinik für Urologie und Kinderurologie der Universität des Saarlandes; Thomas Wiegel, Prof. Dr., Principal Investigator — Klinik für Strahlentherapie und Radioonkologie der Universität Ulm
Locations (2):
- Germany (2):
  - Universitätsklinikum, Ulm, Albert-Einstein-Allee 23
  - Universitätsklinikum, Homburg/Saar, Kirrberger Straße

REFERENCES:
- [Result] Albers P, Wiegel T, Schmidberger H, Bussar-Maatz R, Harter M, Kristiansen G, Martus P, Meisner C, Wellek S, Grozinger K, Renner P, Burmester M, Schneider F, Stockle M. Termination rates and histological reclassification of active surveillance patients with low- and early intermediate-risk prostate cancer: results of the PREFERE trial. World J Urol. 2021 Jan;39(1):65-72. doi: 10.1007/s00345-020-03154-7. Epub 2020 Mar 18. PMID 32189088
- [Result] Wiegel T, Albers P, Bartkowiak D, Bussar-Maatz R, Harter M, Kristiansen G, Martus P, Wellek S, Schmidberger H, Grozinger K, Renner P, Schneider F, Burmester M, Stockle M. Results of a randomized trial of treatment modalities in patients with low or early-intermediate risk prostate cancer (PREFERE trial). J Cancer Res Clin Oncol. 2021 Jan;147(1):235-242. doi: 10.1007/s00432-020-03327-2. Epub 2020 Sep 4. PMID 32886212